CLINICAL TRIAL: NCT07040553
Title: The Effect of an 8-Week Motivational Interviewing and Weekly Digital Messaging Intervention on Premenstrual Symptoms and Emotion Regulation in Female University Students: A Randomized Controlled Trial
Brief Title: Effect of Motivational Interviewing and Digital Support on Premenstrual Symptoms and Emotion Regulation
Acronym: MIND-PMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Collaborators: Erzurum Technical University (Other)
Responsible Party: Principal Investigator, Ayca Balmumcu, Assistant Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ADU-MD-PMS-2025-01; ETU Ethics Committee 2025 (Other: Erzurum Technical University Scientific Research and Publication Ethics Committee)
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Premenstrual Syndrome-PMS; Emotion Regulation
Keywords: Premenstrual Syndrome; Emotion Regulation; Motivational Interviewing; WhatsApp Intervention; Digital Health; University Students; Young Women; Randomized Controlled Trial; Women's health
MeSH Terms: conditions — Premenstrual Syndrome; Emotional Regulation | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Participants were randomized into two parallel groups (intervention and control) using a computer-based algorithm. Group allocation considered participants' residential settings (e.g., dormitory rooms or homes) to minimize intergroup contamination.
Who Masked: Outcomes Assessor
Masking Description: Outcome data were collected by an independent researcher blinded to group allocation to minimize assessment bias
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing and WhatsApp Support (Experimental): Participants in this arm received an 8-week intervention consisting of weekly face-to-face motivational interviews and supportive WhatsApp messages, based on the principles of Motivational Interviewing by Miller and Rollnick (2012).
  Interventions: Behavioral: Motivational Interviewing and WhatsApp Support
- Control Group (No Intervention): Participants in this arm did not receive any intervention during the study period. They completed the same pre- and post-assessments as the experimental group.

INTERVENTIONS:
Behavioral: Motivational Interviewing and WhatsApp Support — This intervention consists of weekly face-to-face motivational interviews and supportive WhatsApp messages, delivered over 8 weeks. It is based on the principles of Motivational Interviewing (Miller & Rollnick, 2012) and aims to support symptom management and emotion regulation in participants with moderate to severe premenstrual syndrome.
  Other Names: Behavioral PMS Support Program
  Arms: Motivational Interviewing and WhatsApp Support

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of an 8-week support program that combines face-to-face motivational interviewing with weekly WhatsApp messages in reducing premenstrual syndrome (PMS) symptoms and improving emotion regulation among university students.

The study was conducted with 70 female students enrolled in the Nursing Department of Erzurum Technical University in Türkiye. Eligible participants are identified using the Premenstrual Syndrome Scale (PMSS), and those scoring above 110 are considered to have PMS. Students who meet the inclusion criteria and volunteer to participate are randomly assigned to either the intervention group (n=35) or the control group (n=35), using a computer-based randomization tool. Housing locations (e.g., dorm rooms or homes) are considered to prevent cross-contamination between groups.

All participants complete three forms: a Personal Information Form (to gather data on sociodemographic, menstrual, and lifestyle characteristics), the PMSS (to assess PMS severity), and the Difficulties in Emotion Regulation Scale - Short Form (DERS-16). These are completed before the intervention and again at 8 weeks.

The intervention group receives weekly one-on-one motivational interviews and supportive WhatsApp messages based on the principles of Motivational Interviewing as defined by Miller and Rollnick (2012). No medical treatments or devices are used in this study. Participation is voluntary, and informed written consent is obtained from all students. Ethical approval was granted by the Ethics Committee of Erzurum Technical University.

DETAILED DESCRIPTION:
This randomized controlled study aims to evaluate the impact of a intervention program on premenstrual syndrome (PMS) symptoms and emotion regulation among female university students in Türkiye. The program includes motivational interviewing and mobile-based support strategies. Participants are selected from nursing students at Erzurum Technical University, based on a set of inclusion criteria such as age, menstrual cycle regularity, and the presence of PMS symptoms above a defined threshold. Individuals with chronic gynecological conditions or recent psychiatric diagnoses are excluded. The minimum required sample size (n = 68) was calculated using G*Power software based on an effect size of 0.76 from Nam and Cha (2019), with α = 0.05 and power = 0.80. To account for potential dropouts and ensure balanced group allocation, a total of 70 eligible participants were recruited and randomly assigned to either the intervention (n = 35) or control (n = 35) group. Data collection tools include the Premenstrual Syndrome Scale (PMSS), the Difficulties in Emotion Regulation Scale - Short Form (DERS-16), and a demographic information form. Ethical approval was obtained from the Ethics Committee of Erzurum Technical University (Decision No: 05/16 - Date: 27.03.2025). Written informed consent was obtained from all participants. The study does not involve the use of any drugs or medical devices.

ELIGIBILITY:
Inclusion Criteria:

* Female university students
* Own and actively use a smartphone with WhatsApp installed
* Have had a regular menstrual cycle (21-35 days) for the past 6 months
* Diagnosed with moderate or severe PMS based on the Premenstrual Syndrome Scale (PMSS)
* Willing to provide written informed consent

Exclusion Criteria:

* Diagnosed with a chronic gynecological condition (e.g., polycystic ovary syndrome, endometriosis)
* Diagnosed with a psychiatric disorder within the past 6 months (e.g., major depression, bipolar disorder, schizophrenia)
* Currently using oral contraceptives
* Currently using medications that may directly affect PMS symptoms (e.g., SSRIs, progesterone-based drugs)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility for participation is based on biological sex assigned at birth due to the study's focus on menstrual cycle-related symptoms (premenstrual syndrome). Gender identity was not a factor in inclusion or exclusion criteria.
Enrollment: 70 (Actual)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Change in Premenstrual Syndrome Severity | Baseline and 8 weeks post-intervention
  Premenstrual Syndrome severity will be measured using the Premenstrual Syndrome Scale (PMSS). Total score change from pre-test to 8 weeks post-intervention will be assessed.

SECONDARY OUTCOMES:
Change in Emotion Regulation | Baseline and 8 weeks post-intervention
  Emotion regulation will be assessed using the Difficulties in Emotion Regulation Scale - Short Form (DERS-16). Score changes between pre- and post-intervention will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Ayça Balmumcu, Assistant Professor, Principal Investigator — Aydin Adnan Menderes University; Nilüfer Yıldırım, Assistant Professor, Study Director — Erzurum Technical University; Semra Elmas, Assistant Professor, Study Director — European University of Lefke
Locations (1):
- Erzurum Technical University, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of individual participant data (IPD) has not yet been determined. Data sharing may be considered following publication of the study results, depending on journal requirements, ethical approvals, and participant confidentiality protections.

REFERENCES:
- [Background] Balmumcu A, Ozturk N. The effect of pilates and a WhatsApp-based health intervention program on symptoms of premenstrual syndrome (PMS): A randomized controlled study. Health Care Women Int. 2024;45(8):929-945. doi: 10.1080/07399332.2023.2294819. Epub 2023 Dec 22. PMID 38133631